CLINICAL TRIAL: NCT03791918
Title: Lenvatinib Plus Programmed Cell Death Protein-1 (PD-1) Antibody Versus Transarterial Chemoembolization for Intermediate-stage Hepatocellular Carcinoma Beyond Up-to-seven Criteria
Brief Title: Lenvatinib Plus PD-1 Antibody vs TACE for Intermediate-stage HCC Beyond Up-to-seven Criteria
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S065
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Lenvatinib; PD-1 Antibody; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; spartalizumab; Pharmaceutical Preparations; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenvatinib Plus PD-1 (Experimental): Participants received lenvatinib capsules 12 milligram (mg) based on the participant's body weight greater than or equal to (>=) 60 kilogram (kg) or 8 mg based on the participant's body weight less than (<) 60 kg at baseline, orally, once daily (QD) in continuous 14-day treatment cycles, and received 3mg/kg PD-1 antibody intravenously every 2 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.
  Interventions: Drug: Lenvatinib; Drug: PD-1 antibody
- TACE (Active Comparator): Hepatic intra-arterial infusion with lipiodol mixed with chemotherapy drugs (EADM, lobaplatin, and MMC), and embolization with polyvinyl alcohol particles (PVA).
  Interventions: Procedure: TACE; Drug: TACE Drug Protocol

INTERVENTIONS:
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
  Other Names: E7080, Lenvima
  Arms: Lenvatinib Plus PD-1
Drug: PD-1 antibody — 3mg/kg intravenously every 2 weeks
  Other Names: Programmed cell death 1 antibody
  Arms: Lenvatinib Plus PD-1
Procedure: TACE — A standard hepatic artery catheter was introduced via the femoral artery percutaneously. Selective catheterization of the proper hepatic artery was performed using standard diagnostic catheters and fluoroscopic guidance. TACE Drug Protocol were injected.
  Other Names: Transarterial chemoembolization
  Arms: TACE
Drug: TACE Drug Protocol — lipiodol mixed with chemotherapy drugs(EADM , lobaplatin, and MMC) followed by polyvinyl alcohol particles (PVA)
  Other Names: Drugs for transarterial chemotherapy and embolization
  Arms: TACE

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lenvatinib combined with PD-1 antibody compared with transarterial chemoembolization (TACE) for patients with intermediate-stage hepatocellular carcinoma (HCC) beyond up-to-seven criteria

DETAILED DESCRIPTION:
Transarterial chemoembolization (TACE) is the most widely used palliative treatment for hepatocellular carcinoma (HCC) patients. While a number of studies demonstrate poor effect of TACE for patients with hepatocellular carcinoma staged BCLC A/B especially for those with tumor beyond up-to-seven criteria. Recently, Lenvatinib was proved non-inferior to sorafenib in overall survival in advanced hepatocellular carcinoma, and Programmed Cell Death Protein-1 (PD-1) antibody was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has evaluated the efficacy and safety of lenvatinib plus PD-1 antibody in intermediate-stage HCC. Thus, the investigators carried out this prospective randomized control to demonstrate the superiority of lenvatinib combined with PD-1 antibody over TACE.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage B
* Beyond up-to-seven criteria (hepatocellular carcinomas with seven as the sum of the size of the largest tumor [in cm] and the number of tumors)
* Eastern Cooperative Oncology Group performance status of 0 to 1
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not applicable for transarterial chemoembolization, surgical resection, and local ablative therapy.
* The following laboratory parameters:

Platelet count ≥ 75,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/ L Serum albumin ≥ 30 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months

SECONDARY OUTCOMES:
Time to progression | 24 months
Adverse Events | 24 months
Progression free survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong